CLINICAL TRIAL: NCT06790407
Title: A Direct-to-Consumer, Randomized, Double-blind, Placebo-controlled Study With Open-label Extension Investigating the Effects of Mimio Biomimetic Cell Care on Metabolic Health in Healthy Overweight Individuals in a Home Setting
Brief Title: Observational Metabolic Health Study
Status: Completed | Type: Observational
Sponsor: Mimio Health, Inc. (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS10
Record Dates: First submitted 2024-12-04; First posted 2025-01-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Healthy Population

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection for NMR lipoprofile, oxidized LDL, hsCRP, HbA1c, Insulin and plasma glucose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mimio Product Group: Participants are randomized to the Mimio Study Product Group or the Placebo.
  Interventions: Dietary Supplement: Mimio Study Product
- Placebo Group: Participants are randomized to the Mimio Study Product Group or the Placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mimio Study Product — Active ingredients in the Mimio study product include Nicotinamide 250mg, Ultra-Micronized Palmitoylethanolamide 600mg, Oleoylethanolamide 400mg, Spermidine 8mg; Other Ingredients: Hydroxypropyl-Methylcellulose (capsule), Silicon Dioxide, Magnesium Stearate.
  Groups: Mimio Product Group
Dietary Supplement: Placebo — Non-active study ingredients in the placebo include Micro Crystalline Cellulose 250mg, Hypromellose, Titanium Dioxide.
  Groups: Placebo Group

SUMMARY:
The rationale for this study is to observe the effect of a consumer-grade commercially available product called Mimio Biomimetic Cell Care on metabolic health in overweight individuals. Additionally, the study aims to observe the effects of the study product on hunger and satiety, as well as effects on cognitive function, sleep, stress, pain, mood, gastrointestinal symptoms and metabolic and inflammatory blood markers via activities that can successfully and effectively be completed in a home setting. Because this product is currently available in the OTC market across the United States, a consumer-driven, decentralized observational clinical research study is well-suited for examining the effects of this study product in this population.

The study will examine outcomes in a broad age range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys, blood sample collection for NMR lipoprofile, oxidized LDL, hsCRP, HbA1c, Insulin and plasma glucose and a saliva sample collection for biological age test. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures, saliva sample collection and blood sample collection at their local laboratory. Findings from this study will contribute knowledge toward the design of future studies and important knowledge on metabolic health.

DETAILED DESCRIPTION:
Intermittent fasting has gained significant scientific and clinical interest in recent years due to its well documented beneficial effects on a wide range of health conditions including cardiovascular disease, metabolic disorders, neurodegenerative conditions, cancer, and autoimmune disease in both clinical and experimental settings. Moreover, prolonged periods of fasting remain one of the only reliable methods of extending lifespan in model organisms due to its reported ability to modulate the cellular aging process. Despite fasting's potential to significantly improve human health by helping to treat, prevent, or delay disease and enhance overall longevity, the prolonged timescale of fasting required to achieve such benefits (typically greater than 24 hrs) is often infeasible or dangerous for numerous populations and adds significant burdens to quality of life which prevent fasting's widespread adoption. Interventions capable of mimicking the beneficial cellular, metabolic, immune, and longevity enhancing effects of fasting without the need to abstain from food, hold great potential therapeutic value for both the treatment and prevention of chronic health conditions especially for those for whom fasting may be contraindicated.

Spermidine, nicotinamide, palmitoylethanolamide (PEA), and oleoylethanolamide (OEA) are endogenous human metabolites that have been shown to have numerous beneficial effects, including improved clinical markers of disease, extended lifespan, and both anti-inflammatory and antioxidant properties. A previous study conducted by the Mimio Health group identified higher plasma concentrations of these metabolites after a 36 hour fast compared to a 12-hour overnight fast and demonstrated that a combination of spermidine, 1-methlynicotinamide (1-MNA): a cellular derivative of nicotinamide, PEA, and OEA could mimic many of the functional benefits of prolonged fasting including significant anti-inflammatory and antioxidant effects in vitro and extending lifespan in C. elegans. The study team has also shown in a pilot clinical study that the combination of spermidine, PEA, OEA, and nicotinamide when taken as a supplement is orally bioavailable, well-tolerated, and capable of replicating similar anti-inflammatory, antioxidant, and cardioprotective effects as fasting even when taken in the postprandial state. The goal of this study is to confirm the beneficial effects of this novel fasting mimetic formulation (Mimio Biomimetic Cell Care) and further explore its potential therapeutic value on metabolic health and longevity in a randomized, double-blind, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years old and above
* Have a BMI between 25 to 29.9 from self-reported weight and height measured within the last 6 months prior to randomization
* Interested in understanding more about their metabolic health
* If taking any prescription medication for cholesterol (e.g. statins) or other class of medications for metabolic disorders such as metformin, ACE inhibitors, beta blockers, rapamycin, thiazolidinediones, etc., must be on a stable dose for at least 4 weeks prior to randomization and throughout the course of the study
* If taking any fiber supplements, must be on a stable dose for at least 4 weeks prior to randomization and throughout the course of the study. If not on a stable dose, must be willing to stop at least 1 week prior to randomization and throughout the course of the study.
* If taking any other supplement products such as fish oil, resveratrol, alpha-ketoglutarate, berberine, ashwagandha, pre- and probiotics, melatonin, NAD+ precursors (niacin, nicotinamide riboside (NR), nicotinamide mononucleotide (NMN), NADH, etc), fisetin, astaxanthin, urolithin-A, CoQ-10, green tea extract or EGG, pterostilbene, must be willing to stop at least 1 week prior to randomization and throughout the course of the study
* If using any cannabis, THC, or CBD containing products regularly, must be willing to stop at least 1 week prior to randomization and throughout the course of the study
* Must be on a consistent and regular diet for at least 2 months prior to randomization and willing to maintain it throughout the course of the study
* For females, must be in menopausal stage
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States.
* Able and willing to travel to a local Quest Diagnostics laboratory for blood sample collection (with fasting) twice during the course of the study
* Able to complete study assessments over the course of up to 10 weeks.

Exclusion Criteria:

-Do not have a personal smartphone, internet access, or unwilling to download Chloe.

Concomitant Therapies:

* GLP-1 receptor agonists and related incretin mimetics, (e.g. semaglutide (Ozempic, Rybelsus), dulaglutide (Trulicity), exenatide (Byetta, Bydureon), liraglutide (Victoza, Saxenda), lixisenatide (Adlyxin), sitagliptin (Januvia, Janumet), saxagliptin (Onglyza, Komblglyze), alogliptin (Nesina, Kazano, Oseni), linagliptin (Tradjenta, Jentadueto) or tirzepatide (Mounjaro))
* Hormone Replacement Therapy (especially fluctuating/ cycle mimicking dose) or Hormonal Contraceptives (oral or IUD)
* Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
* Concurrent participation in any other investigational study during the study period.
* Regular use of over-the-counter allergy or pain medications (including ibuprofen, acetaminophen, aspirin, naproxen, diphenhydramine, cetirizine, loratadine, fexofenadine ) (>3-4 times/week).

Other Illnesses or Conditions: Participants who have the following comorbidities or conditions are excluded:

* Currently or previously diagnosed with Obesity (BMI greater than 29.9)
* Known diagnosis of Type 1 or Type 2 Diabetes Mellitus requiring medical intervention.
* Known diagnosis of an eating disorder
* Currently diagnosed with Alcohol Abuse and/or Substance Use Disorder
* Women not yet in menopause (Have had a menstrual period within the last 12 months)
* Currently diagnosed with Anemia
* Significant cardiovascular disease or severe cardiac event, except hypertension.
* Current or past diagnosis with cancer of any kind, except non-melanoma skin cancer
* Any underlying medical conditions or comorbidities that may confound the evaluation of the study outcomes.
* Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the study or impact the study outcomes.
* Have undergone a major change in diet or on a special diet (e.g. intermittent fasting, carnivore diet, keto diet, vegan/vegetarian, extending fasting etc.) 60 days prior to enrollment or who initiated such a change at any time during the study.
* Recent weight fluctuations (greater than 10% in the last six months)
* Smoker or use of tobacco or nicotine products.
* Regular use of any cannabis, THC, or CBD containing products or unwillingness to cease use of such products 1 week prior to randomization and throughout the duration of the study period.
* Alcohol use exceeding 14 units/week or unwillingness to change drinking habits to 14 or less units/week 1 week prior to randomization and throughout the duration of the study period
* Known hypersensitivity or previous allergic reaction to nicotinamide, palmitoylethanolamide, oleoylethanolamide, spermidine
* Are unlikely for any reason to be able to comply with the trial or considered unsuited for participation in the study by the Principal Investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants who meet the eligibility criteria will be recruited through People Science community, email outreach, advocacy groups and social media channels. Advertisements will be in paper and digital format and will link to a study landing page to enable sign up.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Determine the effect of the study product on hunger and satiety | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  The primary objective of this study is to determine the effect of the study product on hunger and satiety via a 7-item Hunger, Satiety and Cravings scale. The higher the score, the worse the outcome.
  The study team aggregates individual changes in the survey from the baseline period to week 8 and compares placebo and product groups using non-parametric statistics or parametric statistics, depending on final data distribution. Univariate statistics will be generated to describe the distribution of patient characteristics and outcome data. Continuous variables will be described using means, medians, standard deviations/median absolute deviations, minimums and maximums while categorical variables will be described using counts and percentages. The study team is testing the null hypothesis that there is no difference between placebo group and study product groups on mean or ranked scores within study participants.

SECONDARY OUTCOMES:
Assess the effect of the study product on cognitive function | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to assess the effect of Mimio Biomimetic Cell Care product on cognitive function.
  Change in cognitive function as measured by Cognitive Failures Questionnaire (CFQ) score between placebo and study product group. Baseline period will be compared as well.
  The Cognitive Failures Questionnaire (CFQ) is a self-report questionnaire consisting of 25 items assessing deficits regarding attention, perception, memory and motor functioning in everyday life. The total Cognitive Failures Questionnaire score is calculated by summation of all answers and scores range from 0-100. A higher total score indicates more subjective cognitive failure, which is a worse outcome.
Assess the effect of the study product on cognitive and behavioral eating | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to assess the effect of Mimio Biomimetic Cell Care product on cognitive and behavioral components of eating.
  Change in average score on the Three-Factor Eating Questionnaire-r18 between placebo and study product group. Baseline period will be compared as well.
  The Three-Factor Eating Questionnaire-r18 items have four-point response scales ranging from definitely true (score = 4) to definitely false (score = 1). Raw scores are commonly converted into scaled scores of 0-100. Higher scores indicate higher levels of restrained eating, disinhibited eating, and predisposition to hunger, which may indicate a worse outcome.
Assess the effect of the study product on metabolic blood markers | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to assess the effect of Mimio Biomimetic Cell Care product on metabolic blood markers.
  Change from baseline in metabolic blood markers including nuclear magnetic resonance (NMR) lipoprofile, inflammatory marker high-sensitivity C-reactive protein (hsCRP), Hemoglobin A1c (HbA1c), plasma glucose and insulin at Week 8 (End of study) between placebo and study product groups will be analyzed.
  Abnormal bloodwork or significant changes in bloodwork between baseline and end of study will indicate a worse outcome.
Observe the effect of the study product on epigenetic profile/biological age | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to observe the effect of Mimio Biomimetic Cell Care product on epigenetic profile/biological age.
  Change from baseline in the epigenetic profile/biological age between placebo and study product group as measured by the 'TruMe Biological Age Test' at Week 8 (End of study).
  An increase in biological age will indicate a worse outcome.
Assess the effect of the study product on gastrointestinal symptoms | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to assess the effect of Mimio Biomimetic Cell Care product on gastrointestinal symptoms (i.e flatulence, bloating, abdominal discomfort, stool consistency/regularity, constipation.
  Change in average scores of gastrointestinal symptoms (i.e flatulence, bloating, abdominal discomfort, stool consistency/ regularity, constipation) between placebo and study product group as measured by 16 likert scale-type and frequency questions on a weekly survey. Baseline period will be compared as well.
  A higher overall score in weekly gastrointestinal symptoms ratings will indicate worse outcomes.
Assess the effect of the study product on Quality of Life (sleep, stress, mood, energy, and pain) | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to assess the effect of Mimio Biomimetic Cell Care product on quality of life indicators including sleep, stress, mood, energy, and pain.
  Change in average scores on sleep quality, sleep duration, stress, mood, energy and pain between placebo and study product group as measured by 7 likert scale-type and frequency questions on a weekly survey. Baseline period will be compared as well.
  A higher overall score in weekly quality of life ratings will indicate better outcomes.
Observe the effect of the study product on the safety and tolerability | Participants will complete up to a 14-week study consisting of a screening period, randomization and shipping period, a 2-week baseline period, and an 8-week product/placebo use period.
  A secondary objective is to observe the safety and tolerability of Mimio Biomimetic Cell Care product.
  Assessment of the number, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and AE withdrawals reported over the study product/placebo use period.
  A higher number of serious or adverse events will indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided